CLINICAL TRIAL: NCT05110820
Title: Quantitative Assessment of Pupillary Light Reflex for the Prediction of Neurocognitive Outcomes of Acute Carbon Monoxide Poisoning: A Prospective Observational Study
Brief Title: Quantitative Assessment of Pupillary Light Reflex in Acute Carbon Monoxide Poisoning
Status: Completed | Type: Observational
Sponsor: Wonju Severance Christian Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Yong Sung Cha, Assistant Professor, Wonju Severance Christian Hospital
Other Study IDs: CO-pupillometer
Record Dates: First submitted 2021-10-14; First posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Carbon Monoxide Poisoning
MeSH Terms: conditions — Carbon Monoxide Poisoning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute CO poisoning: A diagnosis of CO poisoning was made according to medical history and carboxyhaemoglobin >5% (>10% in smokers).
  Interventions: Diagnostic Test: Automated quantitative pupillometer

INTERVENTIONS:
Diagnostic Test: Automated quantitative pupillometer — Quantitative measurement of pupillary variables was performed at the time of arrival at the ED (0 h), and at the 6-, 12-, and 24-h time points on hospital day (HD) 1. The worst value among those recorded within 24 h and during the total measurement period was selected as the 24-h and total lowest values. If a patient was discharged before HD 3, measurements were taken only until discharge. The initial value was measured within 1 h after arrival at the ED because of the requisite time for obtaining informed consent before enrollment. At each time point, the lowest values for the NPi and qPLR of each eye were retained for analysis. The sPLR (standard PLR) was serially measured in the ED and after admission by emergency physicians using a manual penlight. We classified the reactivity of the sPLR as reactive, sluggish, or non-reactive. Non-reactive sPLR was defined when pupillary reactivity was not identified bilaterally.

SUMMARY:
Neurological complications after acute carbon monoxide (CO) poisoning can range from transient headache or dizziness to cognitive dysfunction, seizure, permanent anoxic brain damages or death. A recent study reported that a lack of standard pupillary light reflex (sPLR), assessed using a pen light, was a predictor of 30-day neurological sequelae in patients with CO poisoning. Given that the basic sPLR has a poor inter-rater reliability, more objective and quantitative methods are required in the assessment of PLR.

An automated pupillometer has been used in the intensive care unit to quantitatively assess the PLR. Therefore, we hypothesized that quantitative assessment of PLR might be associated with neurocognitive sequelae after acute CO poisoning. The purpose of this study was to assess the value of quantitative pupillary reactivity (NPi and qPLR) in comparison to that of sPLR in predicting neurocognitive outcome at 1 month after acute CO poisoning.

DETAILED DESCRIPTION:
Neurological complications after acute carbon monoxide (CO) poisoning can range from transient headache or dizziness to cognitive dysfunction, seizure, permanent anoxic brain damages or death. Although hyperbaric oxygen therapy (HBO2) has been tried to minimize the neurological complications, a significant percentage of patients still suffer from neurocognitive sequelae after acute CO poisoning. A recent study reported that a lack of standard pupillary light reflex (sPLR), assessed using a pen light, was a predictor of 30-day neurological sequelae in patients with CO poisoning. Given that the basic sPLR has a poor inter-rater reliability, more objective and quantitative methods are required in the assessment of PLR.

An automated pupillometer has been used in the intensive care unit to quantitatively assess the PLR. Quantitative PLR (qPLR), which is expressed as the percentage pupillary constriction in response to a calibrated light stimulus, was better in predicting neurological outcome after cardiac arrest (CA) compared to standard light reflex. In addition, the Neurological Pupil index (NPi) has been validated as a tool for assessing prognosis after CA because it is not influenced by medications (especially opioids and neuromuscular blocking agents) or small pupil size.

Therefore, the investigators hypothesized that quantitative assessment of PLR might be associated with neurocognitive sequelae after acute CO poisoning. The purpose of this study was to assess the value of quantitative pupillary reactivity (NPi and qPLR) in comparison to that of sPLR in predicting neurocognitive outcome at 1 month after acute CO poisoning.

ELIGIBILITY:
Inclusion Criteria:

* Acute CO poisoning

Exclusion Criteria:

* Age <19 years
* Patients with a history of ophthalmic surgery which might have affected the PLR
* Patients with baseline cognitive deficit
* Refusal to enroll in this study
* Discharge from the ED or transfer to another hospital within 24 hours
* Expired in the ED
* Co-ingestion of drugs, such as hypnotics, that may affect the PLR
* No follow-up for the neurocognitive outcome

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute CO poisoning
Sampling Method: Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
The prediction of neurological pupil index (NPi) for poor neurocognitive outcome | Within 3 days after acute CO poisoning
  The predictive value of NPi for the 1-month poor neurocognitive outcome after acute CO poisoning
The prediction of quantitative pupillary light reflex (qPLR) for poor neurocognitive outcome | Within 3 days after acute CO poisoning
  The predictive value of qPLR for the 1-month poor neurocognitive outcome after acute CO poisoning
Comparison of predictive value for poor neurocognitive outcome between NPi and standard pupillary light reflex (sPLR) | Within 3 days after acute CO poisoning
  The value of NPi in comparison to that of sPLR in predicting neurocognitive outcome at 1 month after acute CO poisoning
Comparison of predictive value for poor neurocognitive outcome between qPLR and sPLR | Within 3 days after acute CO poisoning
  The value of qPLR in comparison to that of sPLR in predicting neurocognitive outcome at 1 month after acute CO poisoning

CONTACTS AND LOCATIONS:
Locations (1):
- Wonju Severance Christian Hospital, Wŏnju, Gangwon-do, South Korea